CLINICAL TRIAL: NCT04144907
Title: Innovative Approaches to the Lack of Evidence-based Dietary Protein Requirements for Patients With Cancer
Brief Title: Protein Needs Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HREBA.CC-19-0354
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Breast Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phenylalanine intake (Experimental)
  Interventions: Dietary Supplement: Phenylalanine intake

INTERVENTIONS:
Dietary Supplement: Phenylalanine intake — Oral consumption of eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein-free cookies and 4 labeled amino acid experimental meals.

SUMMARY:
Severe muscle loss in patients with cancer has been associated with increased physical disability, extended hospitalization, infectious and noninfectious complications, increased risk of severe toxicity during cancer treatment, poor quality of life and shortened survival. Adequate protein is key to sustain muscle mass and overall health. However, current nutritional recommendations are not specific or evidence-based. The aim of this project is to determine the protein needs of patients with colorectal or breast cancer. Protein needs will be determined using a novel, non-invasive approach. Our results will inform nutritional recommendations and guidelines with the ultimate goal of improving outcomes for people with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients age 45-80 years;
* Patients attending the new patient clinic at the Cross Cancer Institute with a diagnosis of colorectal cancer or breast cancer (stages II to III);
* Able to complete baseline visits within approximately 4 weeks of starting chemotherapy OR after a minimum of 4 weeks post-surgery if not undergoing chemotherapy;
* Ambulatory.

Exclusion Criteria:

* Premenopausal women due to impact on protein requirements;
* Received anti-cancer hormone treatment or immunotherapy in the 4 weeks before first baseline visit;
* Renal impairment based on a creatinine clearance for estimated glomerular filtration rate (eGFR) of <60 mL/min
* Abnormal glucose metabolism based on a fasting glucose level >6mmol/L and an HbA1c >5.7% or as reviewed by study team;
* Comorbidities or medications that would interfere with the participants ability to follow the study protocol or the quality of the data(e.g. diabetes, class III obesity, hormone therapy, another active cancer diagnosis);
* Unable/unwilling to provide urine, breath and blood samples (e.g. oxygen tank, catheter, etc.);
* Unable to eat the meals provided (i.e. receiving parenteral or enteral nutrition, severe allergies);
* Substance dependent (e.g. alcohol, cigarettes, illicit drugs) and unable to follow study protocols.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
13C Phenylalanine Oxidation | 8.5 hours
  Breath, urine and blood samples will be collected during the study to measure the rate of oxidation of 13C phenylalanine.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, RD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No